CLINICAL TRIAL: NCT01857531
Title: Proof-Of-Concept Investigation With a Neurosteroid Analog (Ganaxolone) as a Smoking Cessation Candidate
Acronym: Ganaxolone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jed E. Rose (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Jed E. Rose, Professor, Department of Psychiatry and Behavioral Sciences, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00041533; 1P50DA027840-01A1 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Quit Smoking; Ganaxolone; Nicotine Patch
MeSH Terms: conditions — Smoking Cessation | interventions — ganaxolone; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ganaxolone -- Nicotine Patch (Experimental): Pre-Quit Period:
  Ganaxolone -- 400mg daily for the first 3 days, 800mg daily for the next 3 days and 1200mg daily for the remainder of the first 2 wks.
  Nicotine Patches -- 21mg/24h nicotine patches applied daily during wks. 3 and 4.
  Post-Quit Period:
  Ganaxolone -- 1200mg daily for wk. 5, 800mg daily for 3 days, and 400mg daily for 3 days.
  Nicotine Patches -- 21mg/24h for 4 wks., 14mg/24h for 1 wk., and 7mg/24h for 1 wk.
  Interventions: Drug: Ganaxolone; Drug: Nicotine Patch

INTERVENTIONS:
Drug: Ganaxolone — Pre-Quit Period:
  Beginning at Session P1, subjects will receive ganaxolone at a dose of 400mg total daily (200mg bid) for the first three days, 800mg total daily (400mg bid) for the next three days and 1200mg total daily (600mg bid) for the remainder of the first four weeks.
  Post-Quit Period:
  Following the quit-day, subjects will receive ganaxolone at a dose of (1200mg total daily) for the next week. Down-titration of ganaxolone will begin at post-quit week two. Subjects will receive ganaxolone at a dose of 800mg total daily (400mg bid) to take for three days and 400mg total daily (200mg bid) to take for three.
Drug: Nicotine Patch — Pre-Quit Period:
  Beginning at Session P2, subjects will receive active 21mg/24h nicotine patches to apply daily for the next two weeks.
  Post-Quit Period:
  Following the quit-day, subjects will continue to apply active nicotine patches daily for the remainder of the study (21mg/24h for four weeks, 14mg/24h for one week, and 7mg/24h for one week).
  Other Names: nicoderm

SUMMARY:
The purpose of this research study is to evaluate whether the investigational drug ganaxolone can help smokers quit smoking. Ganaxolone is a drug that has been investigated (in other research studies) for the treatment of seizures and migraines. This drug is considered investigational in the US.

DETAILED DESCRIPTION:
The purpose of this proof-of-concept study is to evaluate whether expired air carbon monoxide (CO) will be reduced and smoking cessation success rates enhanced for smokers who receive the neurosteroid analog ganaxolone. The trial will be seeking preliminary indications of efficacy and tolerability in the smoking population and allow us to estimate effect sizes for future controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Have no known serious medical conditions;
* Are 18-65 years old;
* Smoke an average of at least 10 cigarettes per day;
* Have smoked at least one cumulative year;
* Have an expired air CO reading of at least 10ppm;
* Able to read and understand English;
* Express a desire to quit smoking in the next thirty days.

Potential subjects must agree to use acceptable contraception during their participation in this study.

Potential subjects must agree to avoid the following during their participation in this study:

* participation in any other nicotine-related modification strategy outside of this protocol;
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, e-cigarettes, snuff, and chewing tobacco;
* use of experimental (investigational) drugs or devices;
* use of illegal drugs;
* use of opiate medications;
* consumption of grapefruit or grapefruit juice for the first six weeks of study participation;
* use of melatonin;
* use of sedating antihistamines for the first six weeks of study participation;
* use of alcohol during the first six weeks of study participation.
* use of benzodiazepines

Exclusion Criteria:

* Inability to attend all required experimental sessions;
* Inability to take oral drugs or adhere to medication regimens;
* Hypertension (systolic >140 mm Hg, diastolic >90 mm Hg);
* Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg).
* Coronary heart disease;
* Lifetime history of heart attack;
* Clinically significant cardiac rhythm disorder (irregular heart rhythm);
* Chest pains;
* Cardiac (heart) disorder;
* Extensive active skin disorder;
* Liver or kidney disorder;
* Gastrointestinal disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently symptomatic lung disorder/disease;
* Brain abnormality;
* Migraine headaches that occur more frequently than once per week;
* History of seizures;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes (unless treated with diet and exercise alone);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current symptomatic psychiatric disease;
* Current depression;
* Current suicidal ideation or history of suicide attempt (in the past 5 years);
* Pregnant or nursing mothers;
* Use (within the past 30 days) of:

  * Illegal drugs (or if the urine drug screen is positive),
  * Experimental (investigational) drugs;
  * Psychiatric medications including antidepressants, antipsychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
  * Corticosteroids;
  * Cytochrome P450 341 (CYP3A4) inhibitors and inducers;
  * Smokeless tobacco (chewing tobacco, snuff), pipes or e-cigarettes;
  * Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine replacement therapy or any other smoking cessation aid.
* Use (within the past 14 days) of:

  * dehydroepiandrosterone (DHEA), Pregnenolone or ganaxolone;
  * Opiate medications for pain or sleep;
  * Benzodiazepines or other drugs with significant sedating or anticholinergic activity;
* Use of more than one cigar a month;
* Regular alcohol use;
* Significant adverse reaction to nicotine patches in the past.
* Significant past adverse reaction to ganaxolone in the past.
* Current participation or recent participation (in the past 30 days) in another smoking study at our center or another research facility.
* Current participation in another research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Duke Center for Smoking Cessation, Charlotte, North Carolina
  - Duke Center for Smoking Cessation, Durham, North Carolina
  - Duke Center for Smoking Cessation, Raleigh, North Carolina
  - Duke Center for Smoking Cessation, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Ganaxolone -- Nicotine Patch: Pre-Quit Period:
  Ganaxolone -- 400mg daily (200mg bid) for the first 3 days, 800mg daily (400mg bid) for the next 3 days and 1200mg daily (600mg bid) for the remainder of the first 2 wks.
  Nicotine Patches -- 21mg/24h nicotine patches applied daily during wks. 3 and 4.
  Post-Quit Period:
  Ganaxolone -- 1200mg daily for wk. 5, 800mg daily for 3 days, and 400mg daily for 3 days.
  Nicotine Patches -- 21mg/24h for 4 wks., 14mg/24h for 1 wk., and 7mg/24h for 1 wk.
Period: Overall Study
Arm/Group | Ganaxolone -- Nicotine Patch
Started | 16
Completed | 12
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.44 (9.94)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change in Expired Air Carbon Monoxide (CO) at End of Week 2
Description: To evaluate the effects of ganaxolone on ad lib smoking by looking at the percent change in expired air CO at the end of week two (relative to baseline).
Time Frame: Baseline and 2 Weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 16
percentage change | -0.52 (7.38)

2. Secondary Outcome: Percentage of Change in Expired Air Carbon Monoxide (CO) at End of Week 4
Description: To evaluate the effects of ganaxolone as an augmentation treatment in conjunction with nicotine patch by looking at the percent change in expired air CO at the end of week four (relative to baseline).
Time Frame: Baseline and 4 Weeks
Population: Three of the original 16 subjects dropped out prior to week 4, so only 13 subjects had a week 4 CO reading and could be included in this analysis.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 13
percentage change | -39.40 (8.96)

3. Other Pre Specified Outcome: Number of Participants Completing Continuous 2-week Abstinence From Smoking
Description: Continuous two week abstinence from smoking at the first post-quit visit (approximately 2 weeks post quit date), based on self-reported abstinence confirmed by expired air CO.
Time Frame: 2 Weeks post quit
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 16
participants | 3 [.65 to 7.30]

4. Other Pre Specified Outcome: Number of Participants Completing Point Abstinence From Smoking Two Weeks After Quitting
Description: Point abstinence from smoking two weeks post quit, based on self-reported abstinence during last seven days confirmed by expired air CO at first post-quit visit.
Time Frame: 7 day point abstinence from smoking at 2 weeks post quit
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 16
participants | 4 [1.16 to 8.38]

5. Other Pre Specified Outcome: Number of Participants Completing Continuous 6-week Abstinence From Smoking
Description: Continuous six week abstinence from smoking at final study visit (approximately 6 weeks post quit date), based on self-reported abstinence confirmed by expired air CO
Time Frame: 6 Weeks post quit
Population: Because 6-week abstinence is counted backward from the final study visit, one additional subject (n=4) qualified as abstinent than at 2-weeks post-quit (n=3) due to the fact that the day(s) that one of the subjects smoked did not fall into the range evaluated at 6 weeks.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 16
participants | 4 [1.16 to 8.38]

6. Other Pre Specified Outcome: Number of Participants Completing Abstinence From Smoking During the Last Four Weeks of Treatment
Description: End of treatment abstinence from smoking during the last four weeks of treatment, based on self-reported abstinence during last four weeks confirmed by expired air CO
Time Frame: 4 Week abstinence from smoking at 6 weeks post quit
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Ganaxolone -- Nicotine Patch
Number analyzed (Participants) | 16
participants | 5 [1.76 to 9.39]

ADVERSE EVENTS:
Time Frame: Subjects were receiving study drugs for ten weeks. At each study session during this period subjects completed a questionnaire about side effects. Subjects were also told to contact us between study sessions if side effects were bothersome.
Arm/Group | Ganaxolone -- Nicotine Patch
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ganaxolone -- Nicotine Patch (N=16)
Headache (Nervous system disorders) | 2 (2)
Fatigue (Nervous system disorders) | 11 (15)
Dizziness (Nervous system disorders) | 4 (5)
Loss of balance (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Irritability (Nervous system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (3)
Nightmares (Nervous system disorders) | 1 (1)
Vivid dreams (Nervous system disorders) | 3 (5)
Muscle / joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thirst (General disorders) | 3 (4)
Mouth irritation (General disorders) | 1 (2)
Dry mouth (General disorders) | 1 (1)
Itching at patch site (Skin and subcutaneous tissue disorders) | 5 (7)
Rash at patch site (Skin and subcutaneous tissue disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes